CLINICAL TRIAL: NCT01969617
Title: Interventional, Randomized, Double-blind, Cross-over, Placebo-controlled Study to Investigate the Effects of Nalmefene After Single Dose on the Blood Oxygen Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Signal in the Ventral Striatum to Reward Responding in the Monetary Incentive Delay Task (MIDT), in Non-treatment Seeking Subjects With Alcohol Dependence Following Alcohol Challenge
Brief Title: Effects of Nalmefene After Single Dose on the Blood Oxygen Level Dependent (BOLD) fMRI Signal in the Ventral Striatum to Reward Responding in the Monetary Incentive Delay Task (MIDT), in Non-treatment Seeking Subjects With Alcohol Dependence Following Alcohol Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15660A; 2013-001154-98 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nalmefene 18 mg, then placebo (Experimental): 18 mg nalmefene corresponds to 20 mg nalmefene hydrochloride
  Interventions: Drug: Nalmefene 18 mg, then placebo
- Placebo, then Nalmefene 18 mg (Placebo Comparator): 18 mg nalmefene corresponds to 20 mg nalmefene hydrochloride
  Interventions: Drug: Placebo, then Nalmefene 18 mg

INTERVENTIONS:
Drug: Nalmefene 18 mg, then placebo — One single oral dose Nalmefene on Day 1 and Placebo on Day 8
  Other Names: Selincro®
  Arms: Nalmefene 18 mg, then placebo
Drug: Placebo, then Nalmefene 18 mg — One single oral dose Placebo on Day 1 and Nalmefene on Day 8
  Other Names: Selincro®
  Arms: Placebo, then Nalmefene 18 mg

SUMMARY:
To contribute to the understanding of the underlying neurobiological mechanism behind the interaction of alcohol and nalmefene

ELIGIBILITY:
Inclusion Criteria:

* The subject has alcohol dependence, diagnosed according to DSM-IV-TR™.

Exclusion Criteria:

* The subject is seeking treatment for alcohol dependence.
* The subject has had <6 heavy drinking days (HDDs) in the 4 weeks prior to the Screening Visit.
* The subject has had an average alcohol consumption below high risk levels (that is, 60 grams of alcohol/day for men) <4 weeks prior to the Screening Visit.
* The subject has >5 consecutive abstinence days in the 4 weeks prior to the Screening Visit.
* The subject has a Revised Clinical Institute Withdrawal Assessment of Alcohol Scale, (CIWA-Ar), score ≥10.
* The subject is, in the opinion of the investigator, at significant risk of suicide or meets the exclusion criteria based on C-SSRS.

Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) fMRI signal in the ventral striatum to reward responding using the monetary incentive delay task (MIDT) task | Day 1

SECONDARY OUTCOMES:
Safety | Up to Day 8 and a 10-day safety follow up
  Number of adverse events
Risk of suicidality | Up to Day 8
  Columbia-Suicide Severity Rating Scale (CSSRS) score

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- GB801, London, United Kingdom

REFERENCES:
- [Derived] Quelch DR, Mick I, McGonigle J, Ramos AC, Flechais RSA, Bolstridge M, Rabiner E, Wall MB, Newbould RD, Steiniger-Brach B, van den Berg F, Boyce M, Ostergaard Nilausen D, Breuning Sluth L, Meulien D, von der Goltz C, Nutt D, Lingford-Hughes A. Nalmefene Reduces Reward Anticipation in Alcohol Dependence: An Experimental Functional Magnetic Resonance Imaging Study. Biol Psychiatry. 2017 Jun 1;81(11):941-948. doi: 10.1016/j.biopsych.2016.12.029. Epub 2017 Jan 10. PMID 28216062